CLINICAL TRIAL: NCT04264988
Title: Management and Outcomes of Major Pelvic Hemorrhage in Patients Undergoing Complex Abdomino-Pelvic Surgery: A Cohort Study
Brief Title: Major Pelvic Hemorrhage in Complex Surgery
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Collaborators: Medicana Bursa Hospital (Other); Dokuz Eylul University (Other); Cukurova University (Other); Pamukkale University (Other); Ankara University (Other); TOBB University (Unknown); Gazi University (Other); Baskent University (Other); Ege University (Other); Medipol University (Other); Gulhane Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-6/17
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Pelvic Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who had pelvic hemorrhage: Patients who had pelvic hemorrhage during complex abdomino-pelvic surgery
  Interventions: Procedure: Stopping of pelvic bleeding via several surgical methods

INTERVENTIONS:
Procedure: Stopping of pelvic bleeding via several surgical methods — Those surgical methods were pelvic packing, electrocautery, energy devices, suturing, fastener, muscle welding, procoagulant chemicals, and combination of those

SUMMARY:
Hemorrhage is a challenging complication of pelvic surgery. In this study, the investigators aimed to analyze the causes, management, and outcomes of major pelvic hemorrhage in patients undergoing complex abdomino-pelvic surgery. Participants who had a major intraoperative pelvic hemorrhage during complex abdomino-pelvic surgery at 11 tertiary referral centers were included. Participant characteristics, causes of hemorrhage, management strategies, and outcomes including morbidity and mortality analyses were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had major pelvic bleeding during complex abdominopelvic surgery
* Patients operated in hospitals where over 225 colorectal cases were performed every year

Exclusion Criteria:

* Patients operated for palliative intent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient operated for complex abdominopelvic surgery including radical oncologic operations for the primary advanced or recurrent carcinoma of pelvic organs, pelvic cytoreduction, revisional/redo operations for failed ileal/colonic pouches, repair of the entero-enteral, entero-cutaneous, entero-vesical and entero-vaginal fistulas who had presacral bleeding in centers which had over 225 colorectal cases per year were included. Major pelvic bleeding is defined as symptomatic bleeding originating from pelvis, bleeding leading to transfusion of ≥2 units of whole blood or packed red cells; surgical site bleeding that requires a second intervention; or surgical site bleeding that is unexpected and prolonged and/or sufficiently large to cause hemodynamic instability with an associated decrease in hemoglobin ≥20 g/L.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Peri-operative outcomes | Within postoperative day 30
  Complication rate (Number of participants who had a complication divided by total number of participants)

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Turkey (Türkiye)